CLINICAL TRIAL: NCT03753347
Title: TITRE III: TIV Infant/Toddler Response Evaluation - Influenza B Immunogenicity Investigation
Brief Title: TITRE III: Influenza B Immunogenicity Investigation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: British Columbia Centre for Disease Control (Other Government)
Collaborators: Vaccine Evaluation Center, Canada (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Institut National en Santé Publique du Québec (Other)
Responsible Party: Principal Investigator, Danuta Skowronski, Physician Epidemiologist, Influenza and Emerging Respiratory Pathogens, British Columbia Centre for Disease Control
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H18-02607
Record Dates: First submitted 2018-11-13; First posted 2018-11-27 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- influenza vaccine recipients (Experimental): Participants of an earlier clinical trial (TITRE I) to receive one dose of the 2018-19 quadrivalent inactivated influenza vaccine
  Interventions: Biological: 2018-19 quadrivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: 2018-19 quadrivalent inactivated influenza vaccine — A single age-appropriate dose of 2018-19 quadrivalent inactivated influenza vaccine

SUMMARY:
Each winter, viruses belonging to two kinds of influenza A ("A/H1N1" & "A/H3N2") and two kinds of influenza B ("B/Yamagata" & "B/Victoria") can cause illness. Historically, the yearly influenza vaccine that was recommended in children was designed to protect against both kinds of influenza A but only one kind of influenza B. In a series of trials conducted between 2008-09 and 2010-11 (TITRE I, II, and IIB), the TITRE investigators measured antibody response to influenza B in children who were primed with two doses of trivalent inactivated influenza vaccine (TIV) containing B/Yamagata. Overall, the investigators found that 2 doses of vaccine containing B/Yamagata did not adequately prime children for response to the alternate B/Victoria antigen and that subsequent vaccine doses containing B/Victoria-lineage antigen strongly boosted antibodies to the B/Yamagata antigen that was introduced during first immunization priming, but with lower responses to B/Victoria.

For the first time since 2009-10, the recommended B/Victoria component of the seasonal influenza vaccine has been changed, from B/Brisbane/60/2008 to B/Colorado/60/2007 for the coming 2018-19 season. The investigators thus have a unique opportunity to clarify lineage-specific influenza B responses in a well-characterized cohort of children originally primed to Yamagata. The investigators' main interest is to assess whether TITRE I children primed with two doses of B/Yamagata in 2008-09 have since or are now capable of achieving a sufficient antibody response to B/Victoria following a single dose of 2018-19 QIV, ten years after their initial TIV B/Yamagata priming exposure.

ELIGIBILITY:
Inclusion Criteria:

* Child previously completed the TITRE I study in British Columbia or Quebec;
* Child is healthy (stable chronic conditions acceptable) as established by health assessment interview and verbal history-directed health examination;
* Child is available and can complete all relevant procedures during the study period;
* Parent or legal guardian is available and can be reached by phone during the study period;
* Parent/guardian provides written informed consent;
* Parent/guardian is fluent in English/French

Exclusion Criteria:

* Child has already received the 2018-19 seasonal (TIV or QIV) influenza vaccine;
* Child has a bleeding condition that would prevent vaccine injection or blood collection;
* Child has known or suspected immunodeficiency;
* Child has a suspected or known anaphylactic reaction to any of the vaccine components used in this study;
* Child has a health condition which, in the opinion of the investigator, would interfere with the evaluation or pose a health risk to the child;
* Child has received immune globulin or other blood products within the prior six weeks;
* Child has received injected or oral steroids within the prior six weeks defined by more than 1 week of immunosuppressants or immune modifying drugs (e.g. oral prednisolone >0.5mL/kg/day or intravenous glucocorticoid steroid). Nasal, topical or inhaled steroids are allowed;
* Child has received any live vaccine within 28 days of the study vaccine or is scheduled to receive live vaccine during the study period;
* Child has received any inactivated vaccine within 14 days of the study vaccine;
* Child is or will be enrolled in any other clinical trial of a drug, vaccine or medical device during the study period.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroprotection rate (SPR) for B/Victoria vaccine strains | Pre-vaccination
  SPR based on hemagglutination inhibition (HI) assay for current (B/Colorado/06/2017-like) and prior (B/Brisbane/60/2008-like) Victoria lineage vaccine strains
Seroprotection rate (SPR) for B/Victoria vaccine strains | 4-6 weeks after receipt of QIV
  SPR based on hemagglutination inhibition (HI) assay for current (B/Colorado/06/2017-like) and prior (B/Brisbane/60/2008-like) Victoria lineage vaccine strains

SECONDARY OUTCOMES:
Geometric mean titre (GMT) for B/Victoria vaccine strains | Pre-vaccination
Geometric mean titre (GMT) for B/Victoria vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre ratio (GMTR) for B/Victoria vaccine strains | 4-6 weeks after receipt of QIV
Seroconversion rate (SCR) for B/Victoria vaccine strains | 4-6 weeks after receipt of QIV
Seroprotection rate (SPR) for B/Yamagata vaccine strains | Pre-vaccination
Seroprotection rate (SPR) for B/Yamagata vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre (GMT) for B/Yamagata vaccine strains | Pre-vaccination
Geometric mean titre (GMT) for B/Yamagata vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre ratio (GMTR) for B/Yamagata vaccine strains | 4-6 weeks after receipt of QIV
Seroconversion rate (SCR) for B/Yamagata vaccine strains | 4-6 weeks after receipt of QIV
Seroprotection rate (SPR) for A/H1N1 vaccine strains | Pre-vaccination
Seroprotection rate (SPR) for A/H1N1 vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre (GMT) for A/H1N1 vaccine strains | Pre-vaccination
Geometric mean titre (GMT) for A/H1N1 vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre ratio (GMTR) for A/H1N1 vaccine strains | 4-6 weeks after receipt of QIV
Seroconversion rate (SCR) for A/H1N1 vaccine strains | 4-6 weeks after receipt of QIV
Seroprotection rate (SPR) for A/H3N2 vaccine strains | Pre-vaccination
Seroprotection rate (SPR) for A/H3N2 vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre (GMT) for A/H3N2 vaccine strains | Pre-vaccination
Geometric mean titre (GMT) for A/H3N2 vaccine strains | 4-6 weeks after receipt of QIV
Geometric mean titre ratio (GMTR) for A/H3N2 vaccine strains | 4-6 weeks after receipt of QIV
Seroconversion rate (SCR) for A/H3N2 vaccine strains | 4-6 weeks after receipt of QIV

CONTACTS AND LOCATIONS:
Overall Officials: Danuta M Skowronski, MD, Principal Investigator — BC Centre for Disease Control
Locations (1):
- British Columbia Centre for Disease Control, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Skowronski DM, Hottes TS, De Serres G, Ward BJ, Janjua NZ, Sabaiduc S, Chan T, Petric M. Influenza Beta/Victoria antigen induces strong recall of Beta/Yamagata but lower Beta/Victoria response in children primed with two doses of Beta/Yamagata. Pediatr Infect Dis J. 2011 Oct;30(10):833-9. doi: 10.1097/INF.0b013e31822db4dc. PMID 21857263
- [Background] Skowronski DM, Hottes TS, Chong M, De Serres G, Scheifele DW, Ward BJ, Halperin SA, Janjua NZ, Chan T, Sabaiduc S, Petric M. Randomized controlled trial of dose response to influenza vaccine in children aged 6 to 23 months. Pediatrics. 2011 Aug;128(2):e276-89. doi: 10.1542/peds.2010-2777. Epub 2011 Jul 18. PMID 21768314